CLINICAL TRIAL: NCT01793714
Title: Presurgical Language Mapping With fMRI: Comparison of BOLD and fASL Techniques
Acronym: MALTA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-A00903-40
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Brain Neoplasms
Keywords: Magnetic Resonance Imaging
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

SUMMARY:
One of the aim of the neurosurgical treatment of brain tumor is to offer the maximal resection with the minimal neurological risk. The presurgical mapping of eloquent areas with functional magnetic resonance imaging (fMRI) is helpful to plan the surgery. BOLD fMRI is now the gold standard to map language areas. However, BOLD signal is diminished near the brain tumor. It is now possible to detect cortical activation with arterial spin labeling (ASL) techniques, detecting variations of perfusion during an activation paradigm (fASL), fASL could be interesting to detect eloquent areas near a brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years and older
* Brain tumor involving frontal and/or temporal lobe and/or insula, with scheduled neurosurgery
* Patient able of accepting protocol information
* Patient who received information about the protocol and had not expressed its opposition to participate

Exclusion Criteria:

* Patient with any surgical clip, external clips, or any other ferromagnetic device, that is contraindicated for use in MRI
* Claustrophobic patient
* Patients who cannot cooperate for the fMRI
* Patients subject to major legal protection (safeguarding justice, guardianship, trusteeship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain tumor involving MRI realization
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Qualitative and quantitative comparison of brain activations obtained with both techniques (BOLD fMRI and fASL) | 2 years
  Qualitative and quantitative comparison of brain activations obtained with both techniques (BOLD fMRI and fASL) to presurgically detect language areas located near a brain tumor

SECONDARY OUTCOMES:
Langage laterality index obtained with both techniques (BOLD fMRI and fASL)and fASL) | 2 years
  Size and location of activations obtained with BOLD fMRI and fASL in the presurgical detection of language areas
Difference of cerebral blood flow maps obtained with ASL and fASL | 2 years
  Cerebral blood flow quantification obtained with standard ASL and extracted from fASL

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Ferre, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France